CLINICAL TRIAL: NCT03985982
Title: Randomized Double Blind Phase 3 Study to Assess the Efficacy and Safety of BoNT/A-DP in the Treatment of Glabellar Lines in Comparison With Placebo Followed by an Open Label Extension Study
Brief Title: Botulinum Toxin Treatment of Glabellar Lines: Efficacy and Safety Study III (BLESSIII)
Acronym: BLESSIII
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Croma-Pharma GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CPH-303-201400
Record Dates: First submitted 2019-06-12; First posted 2019-06-14 (Actual); Results first posted 2025-06-05 (Actual); Last update posted 2025-06-05 (Actual); Status verified 2024-12

CONDITIONS: Glabellar Frown Lines
MeSH Terms: interventions — Botulinum Toxins, Type A

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Botulinum toxin A (Experimental): Botulinum Toxin A will be administered in double blind fashion in cycle 1. 20 Units will be administered (divided in five 0.1 mL i.m injections) into glabellar area.
  Interventions: Drug: Botulinum Toxin A
- Placebo (Placebo Comparator): Placebo will be administered in double blind fashion in cycle 1 divided in five 0.1 mL injections into the glabellar area.
  Interventions: Drug: Placebo
- Botulinum toxin A Open Label Extension Arm (Experimental): Open Label Extension Arm where all Subjects from Arm 1 and 2 can receive Experimental Treatment in up to 3 treatment cycles.
  20 Units will be administered (divided in five 0.1 mL i.m. injections) into the glabellar area.
  Interventions: Drug: Botulinum Toxin A

INTERVENTIONS:
Drug: Botulinum Toxin A — Injection, 20 Units divided in five 0.1 mL i.m injections into the glabellar area
  Other Names: BoNT/A-DP
  Arms: Botulinum toxin A
Drug: Placebo — injection, sodium chloride 0.9 % divided in five 0.1 mL i.m injections into the glabellar area
  Other Names: sodium chloride 0,9 %
  Arms: Placebo
Drug: Botulinum Toxin A — Injection, 20 Units divided in five 0.1 mL i.m injections into the glabellar area in up to 3 treatment cycles
  Other Names: BoNT/A-DP
  Arms: Botulinum toxin A Open Label Extension Arm

SUMMARY:
The aim of this study is to assess the efficacy and safety of BoNT/A-DP in the treatment of glabellar lines in comparison with placebo, including efficacy after repeat treatments and long term safety.

DETAILED DESCRIPTION:
The study is a parallel-group, randomized, double blind, placebo-controlled study followed by an open label extension.

An interim Analysis will be performed when all subjects finalized the re-evaluation for retreatment visit at week 16 of the first treatment cycle or completed the double blind phase (whichever occurs earlier).

The first treatment cycle of the study will comprise two treatment groups as follows:

* Group A (active): BoNT/A-DP (20 units, 0.5 mL)
* Group B (placebo control): sterile, 0.9% sodium chloride, (0.5 mL). Eligible subjects will be randomized at baseline (day 0) to Group A or B to receive the first treatment in a 3:1 randomization scheme, respectively. Investigators and subjects will be blinded to the treatment administered and will evaluate the severity of glabellar lines independently. The subject should perform their assessment independently and ideally before the investigator, to ensure they are not biased by the investigator. The same investigator should assess the subject at baseline and at the visits at weeks 1, 2 and 4 in the first treatment cycle.

After a screening period of up to14 calendar days, subjects will receive the first treatment (BoNT/A-DP or placebo) and attend for visits at 1, 2 and 4 weeks after treatment and at 4 weekly intervals thereafter for evaluation of efficacy and safety (primary and key secondary efficacy endpoints are evaluated in the first treatment cycle in comparison with placebo).

The first treatment cycle will last at least 12 weeks and will end when the subjects qualify for re-treatment (in accordance with the "eligibility for re-treatment criteria"). After the first treatment cycle is completed, all subjects may enter the open label extension phase and will be dosed with BoNT/A-DP (20 U) for subsequent re-treatments.

Evaluation for re-treatment takes place at the earliest at 12 weeks after the first/previous treatment. Subjects who do not qualify for re-treatment at week 12 will have the option (pending eligibility) of re-treatment at a later visit (at 4 weekly intervals thereafter) until they are eligible for re-treatment or until a total of 48 weeks has elapsed since study start. Subjects will attend for visits at 1 and 4 weeks after any re-treatment and at 4 weekly intervals thereafter. At week 2 and week 8 of each open label cycle a telephone call visit will take place. According to the study schedule (Section 2.1 and Section 2.2), a maximum of 4 treatments per subject (4 treatment cycles) is permitted during the study time frame, with treatments separated by a minimum of 12 weeks.

The number of treatments administered per subject will depend on the subject's qualification for re-treatment; however, the last opportunity for re-treatment is at week 48.

ELIGIBILITY:
Inclusion Criteria:

* Ages ≥ 18 years or older at time of screening (upper limit 75 years, inclusive).
* Has moderate to severe glabellar frown lines at maximum frown (severity score of 2 or 3 on FWS) as determined by in-clinic assessments by both the investigator and the subject (where: 0 =´none´, 1= ´mild´, 2= ´moderate´, 3= ´severe´).

Subject had a stable medical condition with no uncontrolled systemic disease.

* Female subjects of childbearing potential had to test negative for pregnancy and agree to use effective birth control during the course of the study.
* Subjects who wear glasses had to be able to adequately self-assess the severity of their glabellar lines (according to the FWS), without glasses obstructing the forehead area.
* Moderate to severe glabellar lines indicating an important psychological impact on the subject as indicated by scores > 0 on either the Emotional or the Social Functioning subscale of the Modified Skindex-16 GL-QoL scale.

Exclusion Criteria:

* Previous treatment with any serotype of botulinum toxin for any indication within the 12 months prior to screening, or any planned treatment with botulinum toxin of any serotype for any reason during the study (other than the investigational treatment).
* Known hypersensitivity to the study drug or its excipients.
* Any medical condition that may place the subject at increased risk due to exposure to botulinum toxin, including diagnosed myasthenia gravis, Eaton-Lambert syndrome, amyotrophic lateral sclerosis, profound atrophy or weakness in the target muscles, or any other condition (at the investigator´s discretion) that might interfere with neuromuscular function or contraindicate botulinum toxin therapy.
* Facial laser or light treatment, microdermabrasion, superficial peels or retinoid therapy within the 3 months prior to screening or planned during the study.
* Apart from the procedures specified above, previous treatment with any facial aesthetic procedure in the glabellar area (including chemical peeling, injection with biodegradable fillers) within 12 months prior to screening or planned during the study.
* Previous treatment with any serotype of botulinum toxin for any indication within the 12 months prior to screening, or any planned treatment with botulinum toxin of any serotype for any reason during the trail (other than the investigational treatment).
* Previous insertion of permanent material in the glabellar area or planned during the study.
* Any surgery, or history of surgery, in the glabellar area including surgical removal of the corrugator, procerus or depressor supercilii muscles or a combination of these or scars in the glabellar area or such surgery planned during the study.
* Active skin disease/infection or irritation at the treatment area.
* Inability to substantially lessen glabellar frown lines even by physically spreading them apart.
* Use of a muscle relaxant within 2 weeks prior to screening, or planned during the study.2
* Marked facial asymmetry or ptosis of eyelid and/or eyebrow, or current facial palsy or neuromuscular junction disorders as judged by the investigator.
* Pregnant, breastfeeding or planning to become pregnant during the study.
* Use of prohibited medication including anticholinergic drugs, or drugs that could interfere with neuromuscular function, including aminoglycoside antibiotics and curare-like compounds within 2 weeks prior to screening or planned during the study.2
* Planned surgery with general anesthetic (use of local anesthetic outside the glabellar area was permitted).
* Participation in another clinical study within 1 month of screening and throughout the study.
* Previous participation in another botulinum toxin aesthetic study which involved the treatment of glabellar lines in combination with canthal lines and/or forehead lines, within the previous 18 months.
* Chronic drug or alcohol abuse (as per investigator discretion).

Eligibility Criteria for Retreatment

The following criteria had to be met for retreatment:

* At time of retreatment, the subject did not have relevant changes to their health status from enrolment, which could have prevented the subject's entry into the study according to the inclusion and exclusion criteria.
* The subject had to have been randomized to receive treatment and must have received ≥ 1 treatment (BoNT/A-DP or placebo).
* A minimum of 12 weeks must have elapsed since the previous study treatment.
* The subject's glabellar lines at maximum frown must have relapsed to a FWS score of 2 or 3 as determined by both the investigator and the subject.
* No relevant infection or inflammation in the planned injection area.
* Negative urine pregnancy test, in women of childbearing potential.
* The subject had to have received fewer than 4 study treatments.
* The subject had to have agreed and consented to retreatment.
* Retreatment was to be performed at the latest by Week 48.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 410 (Actual)
Dates: Start 2019-04-29 (Actual); Primary Completion 2019-12-04 (Actual); Study Completion 2020-12-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Adelglass, Dr., Principal Investigator — SKINTASTIC Medical; Sue Ellen Cox, Dr., Principal Investigator — Aesthetic Solutions P.A.; Michael Gold, Dr., Principal Investigator — Tennessee Clinical Research Center; Joely Kaufman-Janette, Dr., Principal Investigator — Skin Research Institute LLC; Susan Taylor, Dr., Principal Investigator — Perelman Center for Advanced Medicine-University of Pennsylvania; Mark Nestor, Dr., Principal Investigator — Center for Clinical and Cosmetic Research; Daniel Mueller, Dr., Principal Investigator — Yuvell (Austria)
Locations (1):
- Tennessee Clinical Research Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No
This is not decided yet and will be changed accordingly when the decision has been made

REFERENCES:
- [Derived] Cox SE, Kaufman-Janette J, Cohen JL, Gold M, Joseph J, Nestor MS, Rzany B, Taylor S, Zhou J, Cecerle M, Pueraro E, Irvine R, Dayan S. LetibotulinumtoxinA Attenuates the Psychological Burden of Glabellar Lines and Is Associated With High Subject Satisfaction in Phase 3 Clinical Trials. Dermatol Surg. 2024 Jun 1;50(6):535-541. doi: 10.1097/DSS.0000000000004152. Epub 2024 Mar 12. PMID 38470985

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of 410 enrolled participants, 355 met inclusion criteria and were randomized to treatment.
Groups:
- Botulinum Toxin A Open Label Extension Arm: Open Label Extension Arm where all Subjects from Arm 1 and 2 can receive Experimental Treatment in up to 3 treatment cycles.
  20 Units will be administered (divided in five 0.1 mL i.m. injections) into the glabellar area.
  Botulinum Toxin A: Injection, 20 Units divided in five 0.1 mL i.m injections into the glabellar area in up to 3 treatment cycles
Period: Double-Blind Phase
Arm/Group | Botulinum Toxin A | Placebo | Botulinum Toxin A Open Label Extension Arm
Started | 266 | 89 | 0
Completed | 250 | 84 | 0
Not Completed | 16 | 5 | 0
Not completed — Lost to Follow-up | 4 | 3 | 0
Not completed — Physician Decision | 1 | 0 | 0
Not completed — Withdrawal by Subject | 9 | 2 | 0
Not completed — COVID-19 | 1 | 0 | 0
Not completed — Early Termination due to Botox Injection while Participating in the Study | 1 | 0 | 0
Period: Open-Label Phase
Arm/Group | Botulinum Toxin A | Placebo | Botulinum Toxin A Open Label Extension Arm
Started | 0 | 0 | 323 (11 participants who completed the Double-Blind Phase did not enroll into the Open-Label Phase because they were not eligible for re-treatment while participating in the study.)
Completed | 0 | 0 | 297
Not Completed | 0 | 0 | 26
Not completed — Lost to Follow-up | 0 | 0 | 13
Not completed — Physician Decision | 0 | 0 | 2
Not completed — Withdrawal by Subject | 0 | 0 | 11

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Botulinum Toxin A | Placebo | Total
Number analyzed (Participants) | 266 | 89 | 355
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 233 | 81 | 314
  >=65 years | 33 | 8 | 41
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.2 (11.24) | 49.4 (12.36) | 51.5 (11.58)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 248 | 80 | 328
  Male | 18 | 9 | 27
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 66 | 22 | 88
  Not Hispanic or Latino | 200 | 67 | 267
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 4 | 1 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 25 | 7 | 32
  White | 236 | 79 | 315
  More than one race | 1 | 2 | 3
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 225 | 79 | 304
  Austria | 41 | 10 | 51
Facial Wrinkle Scale at Maximum Frown by Investigator and Subject In-clinic Assessment [Count of Participants; unit: Participants] — Facial Wrinkle Scale scores are a four-point rating scale as follows: 0 = no facial wrinkles; 1 = mild facial wrinkles; 2 = moderate facial wrinkles; and 3 = severe facial wrinkles.
  Participants
    Investigator's In-clinic Assessment: No facial wrinkles | 0 | 0 | 0
    Investigator's In-clinic Assessment: Mild facial wrinkles | 0 | 0 | 0
    Investigator's In-clinic Assessment: Moderate facial wrinkles | 64 | 22 | 86
    Investigator's In-clinic Assessment: Severe facial wrinkles | 202 | 67 | 269
    Subject's In-clinic Assessment: No facial wrinkles | 0 | 0 | 0
    Subject's In-clinic Assessment: Mild facial wrinkles | 0 | 0 | 0
    Subject's In-clinic Assessment: Moderate facial wrinkles | 70 | 25 | 95
    Subject's In-clinic Assessment: Severe facial wrinkles | 196 | 64 | 260

OUTCOME MEASURES:

1. Primary Outcome: Facial Wrinkle Scale (FWS) Score of 0 or 1 and an Improvement of ≥ 2 Points in FWS Score (at Maximum Frown) at Week 4 Visit Relative to Baseline, Based on Both the Investigators´ and the Subjects´ In-clinic Assessments.
Description: The primary endpoint is the percentage of subjects among BoNT/A-DP and placebo groups with a Facial Wrinkle Scale (FWS) score of 0 or 1 and an improvement of ≥ 2 points in FWS score (at maximum frown) at week 4 visit (of the first treatment cycle) relative to baseline (responders), based on both the investigators' and the subjects' in-clinic assessments. Thus, the primary endpoint is a composite endpoint comprising investigator and subject assessments of treatment effectiveness. FWS scores are a four-point rating scale as follows: 0 = no facial wrinkles; 1 = mild facial wrinkles; 2 = moderate facial wrinkles; and 3 = severe facial wrinkles.
Time Frame: Week 4
Population: The population used consists of all randomized subjects, regardless of whether they received study medication. Participants were analyzed as randomized. Participants with missing investigator or subject in-clinic assessments with the Facial Wrinkle Scale (FWS) at baseline or week 4 were assigned as being non-responders.
Measure: Count of Participants; unit: Participants
Arm/Group | Botulinum Toxin A | Placebo
Number analyzed (Participants) | 266 | 89
Participants | 172 | 0
Statistical Analysis 1: Comparison: Botulinum Toxin A vs Placebo; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel — This outcome measure is the first to be assessed in a hierarchical testing sequence using a one-sided alpha of 0.025

2. Secondary Outcome: Extent of Change in Psychological Impact (Emotional and Social Functioning and Concerns Relating to Glabellar Lines)
Description: Extent of change in psychological impact at week 4 after first treatment, relative to baseline, assessed by
  * modified Skindex-16 (Glabellar Line Quality of Life Scale, [GL-QoL]): Each of 7 items rated on 5-point scale: 0/Never, 1/Rarely, 2/Sometimes, 3/Often, 4/Always bothered, than rescaled to a 0 to 100 standardized score; Emotional Domain is the mean of 4 of the items; Social Functioning Domain is the mean of 3 of the items; Overall score is the mean of all 7 items. All reported scores ranging from 0 (best outcome) to 100 (worst outcome).
  * validated FACE-Q Appraisal of Lines Between Eyebrows scale: Each of 7 items rated on 4-point scale: 1/Not at all, 2/a little, 3/moderately, 4/extremely. Reported score is the sum of the 7 items, standardized on a scale from 0 (worst outcome) to 100 (best outcome).
  * Age Appraisal visual analog scale [VAS]: Perception of Age compared to actual age, in years ranging from -15 years (best outcome) to +15 years (worst outcome).
Time Frame: Week 4
Population: The population used consists of all randomized subjects for whom data are available for the respective timepoint. Participants were analyzed as randomized.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Botulinum Toxin A | Placebo
Number analyzed (Participants) | 264 | 86
score on a scale
  Modified Skindex-16 (GL-QoL) Emotional domain - Change from Baseline at Week 4 | -42.27 (34.484) | 0.50 (20.427)
  Modified Skindex-16 (GL-QoL) Social Functioning domain - Change from Baseline at Week 4 | -33.14 (33.193) | -2.23 (31.088)
  Modified Skindex-16 (GL-QoL) Overall score - Change from Baseline at Week 4 | -38.35 (31.075) | -0.67 (22.369)
  FACE-Q Appraisal of Lines Between Eyebrows - Change from Baseline at Week 4 | 46.4 (28.62) | -2.9 (21.60)
  Age Appraisal VAS - Change from Baseline at Week 4 | -2.3 (4.20) | -0.2 (3.42)
Statistical Analysis 1: Comparison: Botulinum Toxin A vs Placebo; Test performed for Modified Skindex-16 (GL-QoL) Emotional domain - Change from Baseline at Week 4; Test type: Superiority; p < 0.001, Wilcoxon (Mann-Whitney) — The statistical significance is set to 0.025. This is the second test in a hierarchical testing sequence. Statistical significance will only be assessed if the previous test shows statistical significance at the 1-sided alpha level of 0.025
Statistical Analysis 2: Comparison: Botulinum Toxin A vs Placebo; Test performed for Modified Skindex-16 (GL-QoL) Social Functioning domain - Change from Baseline at Week 4; Test type: Superiority; p < 0.001, Wilcoxon (Mann-Whitney) — The statistical significance is set to 0.025. This is the third test in a hierarchical testing sequence. Statistical significance will only be assessed if the previous two tests show statistical significance at the alpha level of 0.025
Statistical Analysis 3: Comparison: Botulinum Toxin A vs Placebo; Test performed for Modified Skindex-16 (GL-QoL) Overall score - Change from Baseline at Week 4; Test type: Superiority; p < 0.001, Wilcoxon (Mann-Whitney) — The statistical significance is set to 0.025. This is the forth test in a hierarchical testing sequence. Statistical significance will only be assessed if the previous three tests show statistical significance at the 1-sided alpha level of 0.025
Statistical Analysis 4: Comparison: Botulinum Toxin A vs Placebo; Test performed for FACE-Q Appraisal of Lines Between Eyebrows - Change from Baseline at Week 4; Test type: Superiority; p < 0.001, Wilcoxon (Mann-Whitney) — The statistical significance is set to 0.025. This is the fifth test in a hierarchical testing sequence. Statistical significance will only be assessed if the previous four tests show statistical significance at the 1-sided alpha level of 0.025
Statistical Analysis 5: Comparison: Botulinum Toxin A vs Placebo; Test performed for FACE-Q Age Appraisal VAS score; Test type: Superiority; p < 0.001, Wilcoxon (Mann-Whitney) — The statistical significance is set to 0.025. This is the sixth test in a hierarchical testing sequence. Statistical significance will only be assessed if the previous five tests show statistical significance at the 1-sided alpha level of 0.025

3. Secondary Outcome: Percentage of Responders at Maximum Frown at Week 12
Description: Percentage of subjects among BoNT/A-DP and placebo groups with a Facial Wrinkle Scale (FWS) score of 0 or 1 and an improvement of ≥ 2 points in FWS score (at maximum frown) at week 12 visit (of the first treatment cycle) relative to baseline (responders), based on both the investigators' and the subjects' in-clinic assessments. FWS scores are a four-point rating scale as follows: 0 = no facial wrinkles; 1 = mild facial wrinkles; 2 = moderate facial wrinkles; and 3 = severe facial wrinkles.
Time Frame: Week 12
Population: The population used consists of all randomized subjects, regardless of whether they received study medication. Participants were analyzed as randomized. Participants with missing investigator or subject in-clinic assessments with the Facial Wrinkle Scale (FWS) at baseline or week 12 were assigned as being non-responders.
Measure: Count of Participants; unit: Participants
Arm/Group | Botulinum Toxin A | Placebo
Number analyzed (Participants) | 266 | 89
Participants | 56 | 1

4. Secondary Outcome: Percentage of Responders at Week 16
Description: Percentage of subjects among BoNT/A-DP and placebo groups with a Facial Wrinkle Scale (FWS) score of 0 or 1 and an improvement of ≥ 2 points in FWS score (at maximum frown) at week 16 visit (of the first treatment cycle) relative to baseline (responders), based on both the investigators' and the subjects' in-clinic assessments. FWS scores are a four-point rating scale as follows: 0 = no facial wrinkles; 1 = mild facial wrinkles; 2 = moderate facial wrinkles; and 3 = severe facial wrinkles.
Time Frame: Week 16
Population: The population used consists of all randomized subjects for whom data are available for week 16 or who were re-treated before week 16. They were analyzed as randomized and participants who were re-treated before week 16 were counted as non-responders.
Measure: Count of Participants; unit: Participants
Arm/Group | Botulinum Toxin A | Placebo
Number analyzed (Participants) | 254 | 84
Participants | 27 | 1

5. Secondary Outcome: Percentage of Responders at Week 20
Description: Percentage of subjects among BoNT/A-DP and placebo groups with a Facial Wrinkle Scale (FWS) score of 0 or 1 and an improvement of ≥ 2 points in FWS score (at maximum frown) at week 20 visit (of the first treatment cycle) relative to baseline (responders), based on both the investigators' and the subjects' in-clinic assessments. FWS scores are a four-point rating scale as follows: 0 = no facial wrinkles; 1 = mild facial wrinkles; 2 = moderate facial wrinkles; and 3 = severe facial wrinkles.
Time Frame: Week 20
Population: The population used consists of all randomized subjects for whom data are available for week 20 or who were re-treated before week 20. They were analyzed as randomized and participants who were re-treated before week 20 were counted as non-responders.
Measure: Count of Participants; unit: Participants
Arm/Group | Botulinum Toxin A | Placebo
Number analyzed (Participants) | 254 | 84
Participants | 5 | 0

6. Secondary Outcome: The Percentage of Subjects With a ≥ 1 Point Reduction in Facial Wrinkle Scale (FWS) Score at Rest at Week 4 Based Separately on the Investigators´ and the Subjects´ In-clinic Assessments
Description: The Percentage of subjects with a ≥ 1 point reduction in Facial Wrinkle Scale (FWS) score at rest at week 4 in the first treatment cycle, based separately on the investigators' and the subjects' in-clinic assessments (applicable only for subjects who have a FWS score at rest ≥ 1 at baseline). FWS scores are a four-point rating scale as follows: 0 = no facial wrinkles; 1 = mild facial wrinkles; 2 = moderate facial wrinkles; and 3 = severe facial wrinkles.
Time Frame: Week 4
Population: The population used consists of all randomized subjects with a Facial Wrinkle Scale (FWS) score at rest >=1 at baseline. Participants were analyzed as randomized. Participants with missing investigator or subject in-clinic assessments with the Facial Wrinkle Scale at week 4 were assigned as being non-responders.
Measure: Count of Participants; unit: Participants
Arm/Group | Botulinum Toxin A | Placebo
Number analyzed (Participants) | 266 | 89
Participants
  Investigator's In-clinic Assessment: number analyzed (Participants) | 215 | 66
  Investigator's In-clinic Assessment | 163 | 8
  Subject's In-clinic Assessment: number analyzed (Participants) | 255 | 82
  Subject's In-clinic Assessment | 214 | 11

7. Secondary Outcome: Responder Rate at Weeks 1, 2 and 8
Description: The Percentage of responders among BoNT/A-DP and placebo groups with a Facial Wrinkle Scale (FWS) score at maximum frown of 0 or 1 and an improvement ≥ 2 points in FWS score (at maximum frown) during the first treatment cycle visit relative to baseline, based on both the investigators' and the subjects' in-clinic assessments (composite endpoint, at weeks 1, 2 and 8). FWS scores are a four-point rating scale as follows: 0 = no facial wrinkles; 1 = mild facial wrinkles; 2 = moderate facial wrinkles; and 3 = severe facial wrinkles.
Time Frame: Week 1, Week 2 and Week 8
Population: The population used consists of all randomized subjects, regardless of whether they received study medication. Participants were analyzed as randomized. Participants with missing investigator or subject in-clinic assessments with the Facial Wrinkle Scale (FWS) at baseline or at the respective visit were assigned as being non-responders.
Measure: Count of Participants; unit: Participants
Arm/Group | Botulinum Toxin A | Placebo
Number analyzed (Participants) | 266 | 89
Participants
  Week 1 | 150 | 0
  Week 2 | 189 | 0
  Week 8 | 129 | 0

8. Secondary Outcome: The Percentage of Subjects With ≥ 2-point and ≥ 1 Reduction in Facial Wrinkle Scale (FWS) Score (at Maximum Frown)
Description: The percentage of subjects with ≥ 2-point and ≥ 1 reduction in Facial Wrinkle Scale (FWS) score (at maximum frown) in the BoNT/A-DP and placebo groups during the first treatment cycle visit relative to baseline, based on the independent rater's assessment of photographs (at baseline and visits 2, 4, 12, 16 and 20 weeks after treatment, within the first treatment cycle). The median value of all assessments of the same photography was considered for analysis. FWS scores are a four-point rating scale as follows: 0 = no facial wrinkles; 1 = mild facial wrinkles; 2 = moderate facial wrinkles; and 3 = severe facial wrinkles.
Time Frame: Week 2, 4, 12, 16 and 20
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Botulinum Toxin A | Placebo
Number analyzed (Participants) | 266 | 89
Participants
  ≥ 2-point reduction - Week 2: number analyzed (Participants) | 256 | 84
  ≥ 2-point reduction - Week 2 | 150 | 0
  ≥ 2-point reduction - Week 4: number analyzed (Participants) | 256 | 85
  ≥ 2-point reduction - Week 4 | 144 | 0
  ≥ 2-point reduction - Week 12: number analyzed (Participants) | 110 | 78
  ≥ 2-point reduction - Week 12 | 11 | 1
  ≥ 2-point reduction - Week 16: number analyzed (Participants) | 55 | 5
  ≥ 2-point reduction - Week 16 | 4 | 0
  ≥ 2-point reduction - Week 20: number analyzed (Participants) | 39 | 1
  ≥ 2-point reduction - Week 20 | 2 | 0
  ≥ 1-point reduction - Week 2: number analyzed (Participants) | 256 | 84
  ≥ 1-point reduction - Week 2 | 235 | 6
  ≥ 1-point reduction - Week 4: number analyzed (Participants) | 256 | 85
  ≥ 1-point reduction - Week 4 | 234 | 9
  ≥ 1-point reduction - Week 12: number analyzed (Participants) | 110 | 78
  ≥ 1-point reduction - Week 12 | 71 | 5
  ≥ 1-point reduction - Week 16: number analyzed (Participants) | 55 | 5
  ≥ 1-point reduction - Week 16 | 29 | 0
  ≥ 1-point reduction - Week 20: number analyzed (Participants) | 39 | 1
  ≥ 1-point reduction - Week 20 | 21 | 1

9. Secondary Outcome: Time to Onset of Effect in the BoNT/A-DP and Placebo Groups in the First Treatment Cycle
Description: Time to onset of effect in the BoNT/A-DP and placebo groups in the first treatment cycle, as measured at weeks 1, 2 and 4 based separately on subject and investigator assessment. Onset of effect defined as at least a 1 point improvement in Facial Wrinkle Scale (FWS) score from baseline (at maximum frown). FWS scores are a four-point rating scale as follows: 0 = no facial wrinkles; 1 = mild facial wrinkles; 2 = moderate facial wrinkles; and 3 = severe facial wrinkles.
Time Frame: From treatment at Day 0 to Week 4 in Treatment Cycle 1
Population: The population used consists of all randomized subjects. Participants were analyzed as randomized.
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | Botulinum Toxin A | Placebo
Number analyzed (Participants) | 266 | 89
Days | 8 [8 to 9] | NA [NA to NA] — The median and inter-quartile range cannot be calculated due to the low number of subjects showing an effect in this arm.

10. Secondary Outcome: Satisfaction With Treatment, During Each Treatment Cycle, as Assessed by the Validated FACE-Q Satisfaction With Outcome Scale.
Description: The extent of subject perceptions of effect of, and satisfaction with, treatment in the BoNT/A-DP and placebo groups, during each treatment cycle, as assessed by the validated FACE-Q Satisfaction with Outcome Scale. The FACE-Q Satisfaction with Outcome scale is a patient-reported outcome measure designed to assess a patient's satisfaction with the results of a facial aesthetic procedure. This scale comprises six items, each with four response options: "definitely agree," "somewhat agree," "somewhat disagree," and "definitely disagree."
Time Frame: Week4 Cycle1(on average 4 Weeks from Baseline, up to Week 7), Week4 Cycle2 (on average 20 Weeks from Baseline, up to Week 52), Week4 Cycle3 (on average 37 Weeks from Baseline, up to Week 53), Week4 Cycle4 (on average 46 Weeks from Baseline, up to Week 56)
Population: The population used consists of all randomized subjects who were treated in the respective study cycle and treatment group. Participants were analyzed as randomized.
Measure: Count of Participants; unit: Participants
Arm/Group | Botulinum Toxin A | Placebo | Botulinum Toxin A Open Label Extension Arm
Number analyzed (Participants) | 266 | 89 | 323
Participants
  Cycle 1 Week 4 - pleased: number analyzed (Participants) | 266 | 89 | 0
  Cycle 1 Week 4 - pleased: Definitely disagree | 16 | 78 |
  Cycle 1 Week 4 - pleased: Somewhat disagree | 13 | 3 |
  Cycle 1 Week 4 - pleased: Somewhat agree | 46 | 4 |
  Cycle 1 Week 4 - pleased: Definitely agree | 189 | 1 |
  Cycle 1 Week 4 - pleased: Missing | 2 | 3 |
  Cycle 1 Week 4 - expected: number analyzed (Participants) | 266 | 89 | 0
  Cycle 1 Week 4 - expected: Definitely disagree | 17 | 74 |
  Cycle 1 Week 4 - expected: Somewhat disagree | 27 | 7 |
  Cycle 1 Week 4 - expected: Somewhat agree | 69 | 5 |
  Cycle 1 Week 4 - expected: Definitely agree | 151 | 0 |
  Cycle 1 Week 4 - expected: Missing | 2 | 3 |
  Cycle 1 Week 4 - great: number analyzed (Participants) | 266 | 89 | 0
  Cycle 1 Week 4 - great: Definitely disagree | 23 | 77 |
  Cycle 1 Week 4 - great: Somewhat disagree | 20 | 7 |
  Cycle 1 Week 4 - great: Somewhat agree | 58 | 2 |
  Cycle 1 Week 4 - great: Definitely agree | 163 | 0 |
  Cycle 1 Week 4 - great: Missing | 2 | 3 |
  Cycle 1 Week 4 - look in the mirror: number analyzed (Participants) | 266 | 89 | 0
  Cycle 1 Week 4 - look in the mirror: Definitely disagree | 18 | 74 |
  Cycle 1 Week 4 - look in the mirror: Somewhat disagree | 34 | 10 |
  Cycle 1 Week 4 - look in the mirror: Somewhat agree | 101 | 2 |
  Cycle 1 Week 4 - look in the mirror: Definitely agree | 111 | 0 |
  Cycle 1 Week 4 - look in the mirror: Missing | 2 | 3 |
  Cycle 1 Week 4 - fantastic: number analyzed (Participants) | 266 | 89 | 0
  Cycle 1 Week 4 - fantastic: Definitely disagree | 25 | 78 |
  Cycle 1 Week 4 - fantastic: Somewhat disagree | 31 | 7 |
  Cycle 1 Week 4 - fantastic: Somewhat agree | 74 | 1 |
  Cycle 1 Week 4 - fantastic: Definitely agree | 134 | 0 |
  Cycle 1 Week 4 - fantastic: Missing | 2 | 3 |
  Cycle 1 Week 4 - miraculous: number analyzed (Participants) | 266 | 89 | 0
  Cycle 1 Week 4 - miraculous: Definitely disagree | 31 | 78 |
  Cycle 1 Week 4 - miraculous: Somewhat disagree | 46 | 8 |
  Cycle 1 Week 4 - miraculous: Somewhat agree | 88 | 0 |
  Cycle 1 Week 4 - miraculous: Definitely agree | 99 | 0 |
  Cycle 1 Week 4 - miraculous: Missing | 2 | 3 |
  Cycle 2 Week 4 - pleased: number analyzed (Participants) | 0 | 0 | 323
  Cycle 2 Week 4 - pleased: Definitely disagree |  |  | 17
  Cycle 2 Week 4 - pleased: Somewhat disagree |  |  | 20
  Cycle 2 Week 4 - pleased: Somewhat agree |  |  | 75
  Cycle 2 Week 4 - pleased: Definitely agree |  |  | 200
  Cycle 2 Week 4 - pleased: Missing |  |  | 11
  Cycle 2 Week 4 - expected: number analyzed (Participants) | 0 | 0 | 323
  Cycle 2 Week 4 - expected: Definitely disagree |  |  | 24
  Cycle 2 Week 4 - expected: Somewhat disagree |  |  | 34
  Cycle 2 Week 4 - expected: Somewhat agree |  |  | 78
  Cycle 2 Week 4 - expected: Definitely agree |  |  | 176
  Cycle 2 Week 4 - expected: Missing |  |  | 11
  Cycle 2 Week 4 - great: number analyzed (Participants) | 0 | 0 | 323
  Cycle 2 Week 4 - great: Definitely disagree |  |  | 30
  Cycle 2 Week 4 - great: Somewhat disagree |  |  | 23
  Cycle 2 Week 4 - great: Somewhat agree |  |  | 80
  Cycle 2 Week 4 - great: Definitely agree |  |  | 179
  Cycle 2 Week 4 - great: Missing |  |  | 11
  Cycle 2 Week 4 - look in the mirror: number analyzed (Participants) | 0 | 0 | 323
  Cycle 2 Week 4 - look in the mirror: Definitely disagree |  |  | 25
  Cycle 2 Week 4 - look in the mirror: Somewhat disagree |  |  | 47
  Cycle 2 Week 4 - look in the mirror: Somewhat agree |  |  | 111
  Cycle 2 Week 4 - look in the mirror: Definitely agree |  |  | 129
  Cycle 2 Week 4 - look in the mirror: Missing |  |  | 11
  Cycle 2 Week 4 - fantastic: number analyzed (Participants) | 0 | 0 | 323
  Cycle 2 Week 4 - fantastic: Definitely disagree |  |  | 36
  Cycle 2 Week 4 - fantastic: Somewhat disagree |  |  | 46
  Cycle 2 Week 4 - fantastic: Somewhat agree |  |  | 90
  Cycle 2 Week 4 - fantastic: Definitely agree |  |  | 140
  Cycle 2 Week 4 - fantastic: Missing |  |  | 11
  Cycle 2 Week 4 - miraculous: number analyzed (Participants) | 0 | 0 | 323
  Cycle 2 Week 4 - miraculous: Definitely disagree |  |  | 52
  Cycle 2 Week 4 - miraculous: Somewhat disagree |  |  | 53
  Cycle 2 Week 4 - miraculous: Somewhat agree |  |  | 105
  Cycle 2 Week 4 - miraculous: Definitely agree |  |  | 102
  Cycle 2 Week 4 - miraculous: Missing |  |  | 11
  Cycle 3 Week 4 - pleased: number analyzed (Participants) | 0 | 0 | 265
  Cycle 3 Week 4 - pleased: Definitely disagree |  |  | 16
  Cycle 3 Week 4 - pleased: Somewhat disagree |  |  | 19
  Cycle 3 Week 4 - pleased: Somewhat agree |  |  | 60
  Cycle 3 Week 4 - pleased: Definitely agree |  |  | 166
  Cycle 3 Week 4 - pleased: Missing |  |  | 4
  Cycle 3 Week 4 - expected: number analyzed (Participants) | 0 | 0 | 265
  Cycle 3 Week 4 - expected: Definitely disagree |  |  | 20
  Cycle 3 Week 4 - expected: Somewhat disagree |  |  | 23
  Cycle 3 Week 4 - expected: Somewhat agree |  |  | 62
  Cycle 3 Week 4 - expected: Definitely agree |  |  | 156
  Cycle 3 Week 4 - expected: Missing |  |  | 4
  Cycle 3 Week 4 - great: number analyzed (Participants) | 0 | 0 | 265
  Cycle 3 Week 4 - great: Definitely disagree |  |  | 24
  Cycle 3 Week 4 - great: Somewhat disagree |  |  | 30
  Cycle 3 Week 4 - great: Somewhat agree |  |  | 56
  Cycle 3 Week 4 - great: Definitely agree |  |  | 151
  Cycle 3 Week 4 - great: Missing |  |  | 4
  Cycle 3 Week 4 - look in the mirror: number analyzed (Participants) | 0 | 0 | 265
  Cycle 3 Week 4 - look in the mirror: Definitely disagree |  |  | 26
  Cycle 3 Week 4 - look in the mirror: Somewhat disagree |  |  | 31
  Cycle 3 Week 4 - look in the mirror: Somewhat agree |  |  | 100
  Cycle 3 Week 4 - look in the mirror: Definitely agree |  |  | 104
  Cycle 3 Week 4 - look in the mirror: Missing |  |  | 4
  Cycle 3 Week 4 - fantastic: number analyzed (Participants) | 0 | 0 | 265
  Cycle 3 Week 4 - fantastic: Definitely disagree |  |  | 35
  Cycle 3 Week 4 - fantastic: Somewhat disagree |  |  | 31
  Cycle 3 Week 4 - fantastic: Somewhat agree |  |  | 72
  Cycle 3 Week 4 - fantastic: Definitely agree |  |  | 123
  Cycle 3 Week 4 - fantastic: Missing |  |  | 4
  Cycle 3 Week 4 - miraculous: number analyzed (Participants) | 0 | 0 | 265
  Cycle 3 Week 4 - miraculous: Definitely disagree |  |  | 52
  Cycle 3 Week 4 - miraculous: Somewhat disagree |  |  | 34
  Cycle 3 Week 4 - miraculous: Somewhat agree |  |  | 77
  Cycle 3 Week 4 - miraculous: Definitely agree |  |  | 98
  Cycle 3 Week 4 - miraculous: Missing |  |  | 4
  Cycle 4 Week 4 - pleased: number analyzed (Participants) | 0 | 0 | 139
  Cycle 4 Week 4 - pleased: Definitely disagree |  |  | 12
  Cycle 4 Week 4 - pleased: Somewhat disagree |  |  | 6
  Cycle 4 Week 4 - pleased: Somewhat agree |  |  | 37
  Cycle 4 Week 4 - pleased: Definitely agree |  |  | 83
  Cycle 4 Week 4 - pleased: Missing |  |  | 1
  Cycle 4 Week 4 - expected: number analyzed (Participants) | 0 | 0 | 139
  Cycle 4 Week 4 - expected: Definitely disagree |  |  | 10
  Cycle 4 Week 4 - expected: Somewhat disagree |  |  | 17
  Cycle 4 Week 4 - expected: Somewhat agree |  |  | 34
  Cycle 4 Week 4 - expected: Definitely agree |  |  | 77
  Cycle 4 Week 4 - expected: Missing |  |  | 1
  Cycle 4 Week 4 - great: number analyzed (Participants) | 0 | 0 | 139
  Cycle 4 Week 4 - great: Definitely disagree |  |  | 17
  Cycle 4 Week 4 - great: Somewhat disagree |  |  | 16
  Cycle 4 Week 4 - great: Somewhat agree |  |  | 33
  Cycle 4 Week 4 - great: Definitely agree |  |  | 72
  Cycle 4 Week 4 - great: Missing |  |  | 1
  Cycle 4 Week 4 - look in the mirror: number analyzed (Participants) | 0 | 0 | 139
  Cycle 4 Week 4 - look in the mirror: Definitely disagree |  |  | 15
  Cycle 4 Week 4 - look in the mirror: Somewhat disagree |  |  | 18
  Cycle 4 Week 4 - look in the mirror: Somewhat agree |  |  | 55
  Cycle 4 Week 4 - look in the mirror: Definitely agree |  |  | 50
  Cycle 4 Week 4 - look in the mirror: Missing |  |  | 1
  Cycle 4 Week 4 - fantastic: number analyzed (Participants) | 0 | 0 | 139
  Cycle 4 Week 4 - fantastic: Definitely disagree |  |  | 21
  Cycle 4 Week 4 - fantastic: Somewhat disagree |  |  | 16
  Cycle 4 Week 4 - fantastic: Somewhat agree |  |  | 46
  Cycle 4 Week 4 - fantastic: Definitely agree |  |  | 55
  Cycle 4 Week 4 - fantastic: Missing |  |  | 1
  Cycle 4 Week 4 - miraculous: number analyzed (Participants) | 0 | 0 | 139
  Cycle 4 Week 4 - miraculous: Definitely disagree |  |  | 29
  Cycle 4 Week 4 - miraculous: Somewhat disagree |  |  | 23
  Cycle 4 Week 4 - miraculous: Somewhat agree |  |  | 45
  Cycle 4 Week 4 - miraculous: Definitely agree |  |  | 41
  Cycle 4 Week 4 - miraculous: Missing |  |  | 1

11. Secondary Outcome: The Percentage of Subjects With a ≥ 1 Point Reduction in Facial Wrinkle Scale (FWS) Score at Rest Based on the Independent Rater's Assessment of Photos.
Description: The percentage of subjects with a ≥ 1 point reduction in Facial Wrinkle Scale (FWS) score at rest in the BoNT/A-DP and placebo groups, relative to baseline, during the first treatment cycle, based on the independent rater's assessment of photos. The median value of all assessments of the same photography was considered for analysis. FWS scores are a four-point rating scale as follows: 0 = no facial wrinkles; 1 = mild facial wrinkles; 2 = moderate facial wrinkles; and 3 = severe facial wrinkles.
Time Frame: Week 2, Week 4, Week 12, Week 16, Week 20 of Treatment Cycle 1
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Botulinum Toxin A | Placebo
Number analyzed (Participants) | 266 | 89
Participants
  Week 2: number analyzed (Participants) | 256 | 84
  Week 2 | 106 | 9
  Week 4: number analyzed (Participants) | 256 | 85
  Week 4 | 100 | 13
  Week 12: number analyzed (Participants) | 110 | 78
  Week 12 | 37 | 8
  Week 16: number analyzed (Participants) | 55 | 5
  Week 16 | 21 | 0
  Week 20: number analyzed (Participants) | 39 | 1
  Week 20 | 11 | 1

12. Secondary Outcome: Facial Wrinkle Scale (FWS) Score of 0 or 1 and an Improvement of ≥ 2 Points in FWS Score (at Maximum Frown) at 4 Weeks After Re-treatment Relative to the Rating at the Preceding End-of-Cycle Visit.
Description: The percentage of subjects with a Facial Wrinkle Scale (FWS) score of 0 or 1 and an improvement of ≥ 2 points in FWS score (at maximum frown) at 4 weeks after re-treatment relative to the rating at the preceding end-of-cycle visit, based on both the investigator's and the subject's in-clinic assessments (composite endpoint). FWS scores are a four-point rating scale as follows: 0 = no facial wrinkles; 1 = mild facial wrinkles; 2 = moderate facial wrinkles; and 3 = severe facial wrinkles.
Time Frame: as for outcome 10
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Botulinum Toxin A Open Label Extension Arm
Number analyzed (Participants) | 323
Participants
  Week 4 after 1st Re-treatment: number analyzed (Participants) | 312
  Week 4 after 1st Re-treatment | 153
  Week 4 after 2nd Re-treatment: number analyzed (Participants) | 253
  Week 4 after 2nd Re-treatment | 119
  Week 4 after 3rd Re-treatment: number analyzed (Participants) | 138
  Week 4 after 3rd Re-treatment | 43

13. Secondary Outcome: The Percentage of Subjects With ≥ 1-point Reduction in Facial Wrinkle Scale (FWS) Score (at Maximum Frown) During the First Treatment Cycle at Week 1, 2, 4, 8, 12, 16 and 20 Relative to Baseline
Description: The percentage of subjects with ≥ 1-point reduction in Facial Wrinkle Scale (FWS) score (at maximum frown) in the BoNT/A-DP and placebo groups during the first treatment cycle at week 1, 2, 4, 8, 12, 16 and 20 relative to baseline, based on both the investigators' and the subjects' in-clinic assessments (composite endpoint). For week 16 and 20 subjects who were re-treated before the respective visits were counted as non-responders. FWS scores are a four-point rating scale as follows: 0 = no facial wrinkles; 1 = mild facial wrinkles; 2 = moderate facial wrinkles; and 3 = severe facial wrinkles.
Time Frame: Week 1, Week 2, Week 4, Week 8, Week 12, Week 16, Week 20 of Treatment Cycle 1
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Botulinum Toxin A | Placebo
Number analyzed (Participants) | 266 | 89
Participants
  Week 1 | 220 | 2
  Week 2 | 234 | 0
  Week 4 | 236 | 0
  Week 8 | 213 | 1
  Week 12 | 162 | 2
  Week 16: number analyzed (Participants) | 254 | 84
  Week 16 | 94 | 1
  Week 20: number analyzed (Participants) | 254 | 84
  Week 20 | 46 | 0

14. Secondary Outcome: The Percentage of Subjects With ≥ 1-point Reduction in Facial Wrinkle Scale (FWS) Score (at Maximum Frown) During Each Re-treatment Cycle at Week 4 Relative to Re-treatment-baseline.
Description: The percentage of subjects with ≥ 1-point reduction in Facial Wrinkle Scale (FWS) score (at maximum frown) in the BoNT/A-DP during each re-treatment cycle at week 4 relative to re-treatment baseline, based on both the investigators' and the subjects' in-clinic assessments (composite endpoint). FWS scores are a four-point rating scale as follows: 0 = no facial wrinkles; 1 = mild facial wrinkles; 2 = moderate facial wrinkles; and 3 = severe facial wrinkles.
Time Frame: as for outcome 10
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Botulinum Toxin A Open Label Extension Arm
Number analyzed (Participants) | 323
Participants
  Week 4 after 1st Re-treatment: number analyzed (Participants) | 312
  Week 4 after 1st Re-treatment | 267
  Week 4 after 2nd Re-treatment: number analyzed (Participants) | 253
  Week 4 after 2nd Re-treatment | 210
  Week 4 after 3rd Re-treatment: number analyzed (Participants) | 138
  Week 4 after 3rd Re-treatment | 104

15. Secondary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs), Serious AEs (SAEs) and AEs of Special Interest (AESIs)
Description: Number of Participants with treatment-emergent adverse events (TEAEs), serious AEs (SAEs) and AEs of special interest (AESIs)
Time Frame: Through study completion (60 weeks)
Population: The population used consists of all subjects who received at least one injection with study medication. Participants were analyzed as treated.
Measure: Count of Participants; unit: Participants
Arm/Group | Botulinum Toxin A | Placebo | Botulinum Toxin A Open Label Extension Arm
Number analyzed (Participants) | 266 | 89 | 323
Participants
  Subjects with any Treatment Emergent Adverse Event (TEAE) | 48 | 14 | 80
  Subjects with any Study Medication Related TEAE | 4 | 0 | 8
  Subjects with any Injection Procedure Related TEAE | 4 | 0 | 6
  Subjects with any Severe TEAE | 1 | 0 | 3
  Subjects with severe study drug related TEAE | 0 | 0 | 0
  Subjects with severe injection procedure related TEAE | 0 | 0 | 0
  Subjects with any Serious TEAE | 1 | 1 | 4
  Subjects with any Adverse Events of Special Interest (AESI) | 1 | 0 | 7
  Subjects with any TEAE leading to discontinuation | 0 | 0 | 0

16. Secondary Outcome: Number of Participants With Neutralizing Anti-Drug Antibodies
Description: Number of Participants with Neutralizing Anti-Drug Antibodies Antibody formation, evaluation pre-dose before each treatment, at 4 weeks after each treatment and at the final study visit.
Time Frame: Through study completion (60 weeks)
Population: The population used consists of all subjects who received at least one injection with study medication. Participants were analyzed as treated. Confirmation assays have only been performed for subjects with a reactive Screening Assay result.
Measure: Count of Participants; unit: Participants
Arm/Group | Botulinum Toxin A | Placebo | Botulinum Toxin A Open Label Extension Arm
Number analyzed (Participants) | 266 | 89 | 323
Participants
  Baseline - Anti-Drug Antibodies (ADA) Screening Assay - Reactive: number analyzed (Participants) | 266 | 89 | 0
  Baseline - Anti-Drug Antibodies (ADA) Screening Assay - Reactive | 23 | 4 |
  Baseline - ADA Confirmation Assay - Confirmed: number analyzed (Participants) | 23 | 4 | 0
  Baseline - ADA Confirmation Assay - Confirmed | 0 | 0 |
  End of Study - ADA Screening Assay - Reactive: number analyzed (Participants) | 0 | 0 | 250
  End of Study - ADA Screening Assay - Reactive | 0 | 0 | 21
  End of Study - ADA Confirmation Assay - Confirmed: number analyzed (Participants) | 0 | 0 | 21
  End of Study - ADA Confirmation Assay - Confirmed | 0 | 0 | 0

17. Secondary Outcome: Change From Baseline of Basophils, Eosinophils, Leukocytes, Lymphocytes, Monocytes, Neutrophils, Platelets
Description: Safety assessments by evaluating change from baseline of Basophils, Eosinophils, Leukocytes, Lymphocytes, Monocytes, Neutrophils, Platelets as per the study schedule
Time Frame: as for outcome 10
Population: The population used consists of all subjects who received at least one injection with study medication and have data available for the respective visit. Participants were analyzed as treated.
Measure: Mean (Standard Deviation); unit: x10^9 cells/L
Groups:
- Botulinum Toxin A: Botulinum Toxin A will be administered in double blind fashion in Treatment Cycle 1. 20 Units will be administered (divided in five 0.1 mL i.m injections) into glabellar area.
  Botulinum Toxin A: Injection, 20 Units divided in five 0.1 mL i.m injections into the glabellar area
- Placebo: Placebo will be administered in double blind fashion in Treatment Cycle 1 divided in five 0.1 mL injections into the glabellar area.
  Placebo: injection, sodium chloride 0.9 % divided in five 0.1 mL i.m injections into the glabellar area
- Botulinum Toxin A Open Label Extension Arm: Open Label Extension Arm where all Subjects from Arm 1 (Botulin toxin A) and 2 (Placebo) can receive Experimental Treatment in up to three additional treatment cycles (cycle 2, 3 and 4).
  Botulinum Toxin A: Injection, 20 Units divided in five 0.1 mL i.m injections into the glabellar area
Arm/Group | Botulinum Toxin A | Placebo | Botulinum Toxin A Open Label Extension Arm
Number analyzed (Participants) | 250 | 82 | 299
x10^9 cells/L
  Week 4 of cycle 1 - Basophils (x10^9 cells/L): number analyzed (Participants) | 250 | 82 | 0
  Week 4 of cycle 1 - Basophils (x10^9 cells/L) | 0.004 (0.0413) | 0.012 (0.0556) |
  Week 4 of cycle 1 - Eosinophils (x10^9 cells/L): number analyzed (Participants) | 250 | 82 | 0
  Week 4 of cycle 1 - Eosinophils (x10^9 cells/L) | 0.006 (0.0726) | 0.007 (0.0767) |
  Week 4 of cycle 1 - Leukocytes (x10^9 cells/L): number analyzed (Participants) | 250 | 82 | 0
  Week 4 of cycle 1 - Leukocytes (x10^9 cells/L) | -0.029 (1.4925) | 0.227 (1.4308) |
  Week 4 of cycle 1 - Lymphocytes (x10^9 cells/L): number analyzed (Participants) | 250 | 82 | 0
  Week 4 of cycle 1 - Lymphocytes (x10^9 cells/L) | -0.038 (0.4554) | -0.027 (0.4222) |
  Week 4 of cycle 1 - Monocytes (x10^9 cells/L): number analyzed (Participants) | 250 | 82 | 0
  Week 4 of cycle 1 - Monocytes (x10^9 cells/L) | -0.027 (0.1607) | -0.019 (0.2154) |
  Week 4 of cycle 1 - Neutrophils (x10^9 cells/L): number analyzed (Participants) | 250 | 82 | 0
  Week 4 of cycle 1 - Neutrophils (x10^9 cells/L) | 0.027 (1.3211) | 0.252 (1.1477) |
  Week 4 of cycle 1 - Platelets (x10^9 cells/L): number analyzed (Participants) | 250 | 80 | 0
  Week 4 of cycle 1 - Platelets (x10^9 cells/L) | 0.3 (37.31) | -0.8 (38.87) |
  Week 4 of cycle 2 - Basophils (x10^9 cells/L): number analyzed (Participants) | 0 | 0 | 299
  Week 4 of cycle 2 - Basophils (x10^9 cells/L) |  |  | -0.002 (0.0565)
  Week 4 of cycle 2 - Eosinophils (x10^9 cells/L): number analyzed (Participants) | 0 | 0 | 299
  Week 4 of cycle 2 - Eosinophils (x10^9 cells/L) |  |  | 0.009 (0.0998)
  Week 4 of cycle 2 - Leukocytes (x10^9 cells/L): number analyzed (Participants) | 0 | 0 | 299
  Week 4 of cycle 2 - Leukocytes (x10^9 cells/L) |  |  | 0.000 (1.5182)
  Week 4 of cycle 2 - Lymphocytes (x10^9 cells/L): number analyzed (Participants) | 0 | 0 | 299
  Week 4 of cycle 2 - Lymphocytes (x10^9 cells/L) |  |  | 0.043 (0.4282)
  Week 4 of cycle 2 - Monocytes (x10^9 cells/L): number analyzed (Participants) | 0 | 0 | 299
  Week 4 of cycle 2 - Monocytes (x10^9 cells/L) |  |  | -0.002 (0.1123)
  Week 4 of cycle 2 - Neutrophils (x10^9 cells/L): number analyzed (Participants) | 0 | 0 | 299
  Week 4 of cycle 2 - Neutrophils (x10^9 cells/L) |  |  | -0.048 (1.3470)
  Week 4 of cycle 2 - Platelets (x10^9 cells/L): number analyzed (Participants) | 0 | 0 | 299
  Week 4 of cycle 2 - Platelets (x10^9 cells/L) |  |  | 6.1 (37.89)
  Week 4 of cycle 3 - Basophils (x10^9 cells/L): number analyzed (Participants) | 0 | 0 | 234
  Week 4 of cycle 3 - Basophils (x10^9 cells/L) |  |  | -0.018 (0.0496)
  Week 4 of cycle 3 - Eosinophils (x10^9 cells/L): number analyzed (Participants) | 0 | 0 | 234
  Week 4 of cycle 3 - Eosinophils (x10^9 cells/L) |  |  | -0.002 (0.1059)
  Week 4 of cycle 3 - Leukocytes (x10^9 cells/L): number analyzed (Participants) | 0 | 0 | 234
  Week 4 of cycle 3 - Leukocytes (x10^9 cells/L) |  |  | -0.050 (2.0753)
  Week 4 of cycle 3 - Lymphocytes (x10^9 cells/L): number analyzed (Participants) | 0 | 0 | 234
  Week 4 of cycle 3 - Lymphocytes (x10^9 cells/L) |  |  | 0.021 (0.4473)
  Week 4 of cycle 3 - Monocytes (x10^9 cells/L): number analyzed (Participants) | 0 | 0 | 234
  Week 4 of cycle 3 - Monocytes (x10^9 cells/L) |  |  | -0.018 (0.1246)
  Week 4 of cycle 3 - Neutrophils (x10^9 cells/L): number analyzed (Participants) | 0 | 0 | 234
  Week 4 of cycle 3 - Neutrophils (x10^9 cells/L) |  |  | -0.034 (1.9383)
  Week 4 of cycle 3 - Platelets (x10^9 cells/L): number analyzed (Participants) | 0 | 0 | 233
  Week 4 of cycle 3 - Platelets (x10^9 cells/L) |  |  | 6.1 (39.16)
  Week 4 of cycle 4 - Basophils (x10^9 cells/L): number analyzed (Participants) | 0 | 0 | 126
  Week 4 of cycle 4 - Basophils (x10^9 cells/L) |  |  | -0.019 (0.0475)
  Week 4 of cycle 4 - Eosinophils (x10^9 cells/L): number analyzed (Participants) | 0 | 0 | 126
  Week 4 of cycle 4 - Eosinophils (x10^9 cells/L) |  |  | -0.026 (0.0859)
  Week 4 of cycle 4 - Leukocytes (x10^9 cells/L): number analyzed (Participants) | 0 | 0 | 126
  Week 4 of cycle 4 - Leukocytes (x10^9 cells/L) |  |  | -0.404 (1.5800)
  Week 4 of cycle 4 - Lymphocytes (x10^9 cells/L): number analyzed (Participants) | 0 | 0 | 126
  Week 4 of cycle 4 - Lymphocytes (x10^9 cells/L) |  |  | 0.003 (0.4665)
  Week 4 of cycle 4 - Monocytes (x10^9 cells/L): number analyzed (Participants) | 0 | 0 | 126
  Week 4 of cycle 4 - Monocytes (x10^9 cells/L) |  |  | -0.025 (0.1698)
  Week 4 of cycle 4 - Neutrophils (x10^9 cells/L): number analyzed (Participants) | 0 | 0 | 126
  Week 4 of cycle 4 - Neutrophils (x10^9 cells/L) |  |  | -0.344 (1.3644)
  Week 4 of cycle 4 - Platelets (x10^9 cells/L): number analyzed (Participants) | 0 | 0 | 126
  Week 4 of cycle 4 - Platelets (x10^9 cells/L) |  |  | 0.4 (41.64)

18. Secondary Outcome: Change From Baseline of Alanine Aminotransferase, Alkaline Phosphatase , Aspartate Aminotransferase, Gamma Glutamyl Transpeptidase
Description: Safety assessments by evaluating change from baseline of Alanine Aminotransferase, Alkaline Phosphatase , Aspartate Aminotransferase, Gamma Glutamyl Transpeptidase as per the study schedule
Time Frame: as for outcome 10
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Botulinum Toxin A | Placebo | Botulinum Toxin A Open Label Extension Arm
Number analyzed (Participants) | 259 | 84 | 301
U/L
  Week 4 of cycle 1 - Alanine Aminotransferase (U/L): number analyzed (Participants) | 254 | 82 | 0
  Week 4 of cycle 1 - Alanine Aminotransferase (U/L) | -0.1 (9.32) | 1.9 (19.35) |
  Week 4 of cycle 1 - Alkaline phosphatase (U/L): number analyzed (Participants) | 259 | 84 | 0
  Week 4 of cycle 1 - Alkaline phosphatase (U/L) | -0.8 (10.99) | -0.5 (12.30) |
  Week 4 of cycle 1 - Aspartate Aminotransferase (U/L): number analyzed (Participants) | 254 | 82 | 0
  Week 4 of cycle 1 - Aspartate Aminotransferase (U/L) | 0.2 (11.28) | 0.1 (8.63) |
  Week 4 of cycle 1 - Gamma Glutamyl Transpeptidase (U/L): number analyzed (Participants) | 259 | 84 | 0
  Week 4 of cycle 1 - Gamma Glutamyl Transpeptidase (U/L) | 0.8 (50.89) | 0.8 (12.41) |
  Week 4 of cycle 2 - Alanine Aminotransferase (U/L): number analyzed (Participants) | 0 | 0 | 300
  Week 4 of cycle 2 - Alanine Aminotransferase (U/L) |  |  | 1.1 (10.68)
  Week 4 of cycle 2 - Alkaline phosphatase (U/L): number analyzed (Participants) | 0 | 0 | 301
  Week 4 of cycle 2 - Alkaline phosphatase (U/L) |  |  | 0.9 (9.42)
  Week 4 of cycle 2 - Aspartate Aminotransferase (U/L): number analyzed (Participants) | 0 | 0 | 301
  Week 4 of cycle 2 - Aspartate Aminotransferase (U/L) |  |  | -0.2 (12.76)
  Week 4 of cycle 2 - Gamma Glutamyl Transpeptidase (U/L): number analyzed (Participants) | 0 | 0 | 301
  Week 4 of cycle 2 - Gamma Glutamyl Transpeptidase (U/L) |  |  | 1.3 (11.09)
  Week 4 of cycle 3 - Alanine Aminotransferase (U/L): number analyzed (Participants) | 0 | 0 | 233
  Week 4 of cycle 3 - Alanine Aminotransferase (U/L) |  |  | -0.4 (13.43)
  Week 4 of cycle 3 - Alkaline phosphatase (U/L): number analyzed (Participants) | 0 | 0 | 234
  Week 4 of cycle 3 - Alkaline phosphatase (U/L) |  |  | 0.6 (10.89)
  Week 4 of cycle 3 - Aspartate Aminotransferase (U/L): number analyzed (Participants) | 0 | 0 | 233
  Week 4 of cycle 3 - Aspartate Aminotransferase (U/L) |  |  | -1.0 (14.73)
  Week 4 of cycle 3 - Gamma Glutamyl Transpeptidase (U/L): number analyzed (Participants) | 0 | 0 | 234
  Week 4 of cycle 3 - Gamma Glutamyl Transpeptidase (U/L) |  |  | 0.0 (9.64)
  Week 4 of cycle 4 - Alanine Aminotransferase (U/L): number analyzed (Participants) | 0 | 0 | 127
  Week 4 of cycle 4 - Alanine Aminotransferase (U/L) |  |  | -0.2 (10.82)
  Week 4 of cycle 4 - Alkaline phosphatase (U/L): number analyzed (Participants) | 0 | 0 | 127
  Week 4 of cycle 4 - Alkaline phosphatase (U/L) |  |  | 0.9 (10.75)
  Week 4 of cycle 4 - Aspartate Aminotransferase (U/L): number analyzed (Participants) | 0 | 0 | 127
  Week 4 of cycle 4 - Aspartate Aminotransferase (U/L) |  |  | -1.6 (14.54)
  Week 4 of cycle 4 - Gamma Glutamyl Transpeptidase (U/L): number analyzed (Participants) | 0 | 0 | 127
  Week 4 of cycle 4 - Gamma Glutamyl Transpeptidase (U/L) |  |  | 1.0 (9.59)

19. Secondary Outcome: Change From Baseline of Cholesterol, Glucose, Potassium, Sodium, Urea Nitrogen
Description: Safety assessments by evaluating change from baseline of Cholesterol, Glucose, Potassium, Sodium, Urea Nitrogen as per the study schedule
Time Frame: as for outcome 10
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Botulinum Toxin A | Placebo | Botulinum Toxin A Open Label Extension Arm
Number analyzed (Participants) | 259 | 84 | 301
mmol/L
  Week 4 of cycle 1 - Cholesterol (mmol/L): number analyzed (Participants) | 259 | 84 | 0
  Week 4 of cycle 1 - Cholesterol (mmol/L) | -0.119 (0.6477) | -0.049 (0.5400) |
  Week 4 of of cycle 1 - Glucose (mmol/L): number analyzed (Participants) | 255 | 82 | 0
  Week 4 of of cycle 1 - Glucose (mmol/L) | 0.317 (1.1751) | 0.290 (0.9429) |
  Week 4 of of cycle 1 - Potassium (mmol/L): number analyzed (Participants) | 259 | 84 | 0
  Week 4 of of cycle 1 - Potassium (mmol/L) | -0.06 (0.405) | -0.09 (0.431) |
  Week 4 of of cycle 1 - Sodium (mmol/L): number analyzed (Participants) | 259 | 84 | 0
  Week 4 of of cycle 1 - Sodium (mmol/L) | -0.1 (2.39) | -0.3 (2.35) |
  Week 4 of of cycle 1 - Urea nitrogen (mmol/L): number analyzed (Participants) | 259 | 84 | 0
  Week 4 of of cycle 1 - Urea nitrogen (mmol/L) | 0.01 (1.356) | 0.00 (1.123) |
  Week 4 of cycle 2 - Cholesterol (mmol/L): number analyzed (Participants) | 0 | 0 | 301
  Week 4 of cycle 2 - Cholesterol (mmol/L) |  |  | 0.07 (0.5910)
  Week 4 of of cycle 2 - Glucose (mmol/L): number analyzed (Participants) | 0 | 0 | 301
  Week 4 of of cycle 2 - Glucose (mmol/L) |  |  | 0.086 (1.2927)
  Week 4 of of cycle 2 - Potassium (mmol/L): number analyzed (Participants) | 0 | 0 | 301
  Week 4 of of cycle 2 - Potassium (mmol/L) |  |  | 0.03 (0.391)
  Week 4 of of cycle 2 - Sodium (mmol/L): number analyzed (Participants) | 0 | 0 | 301
  Week 4 of of cycle 2 - Sodium (mmol/L) |  |  | -0.1 (2.28)
  Week 4 of of cycle 2 - Urea nitrogen (mmol/L): number analyzed (Participants) | 0 | 0 | 301
  Week 4 of of cycle 2 - Urea nitrogen (mmol/L) |  |  | -0.05 (1.277)
  Week 4 of cycle 3 - Cholesterol (mmol/L): number analyzed (Participants) | 0 | 0 | 234
  Week 4 of cycle 3 - Cholesterol (mmol/L) |  |  | 0.021 (0.7421)
  Week 4 of of cycle 3 - Glucose (mmol/L): number analyzed (Participants) | 0 | 0 | 234
  Week 4 of of cycle 3 - Glucose (mmol/L) |  |  | 0.185 (1.5644)
  Week 4 of of cycle 3 - Potassium (mmol/L): number analyzed (Participants) | 0 | 0 | 234
  Week 4 of of cycle 3 - Potassium (mmol/L) |  |  | 0.03 (0.415)
  Week 4 of of cycle 3 - Sodium (mmol/L): number analyzed (Participants) | 0 | 0 | 234
  Week 4 of of cycle 3 - Sodium (mmol/L) |  |  | 0.1 (2.44)
  Week 4 of of cycle 3 - Urea nitrogen (mmol/L): number analyzed (Participants) | 0 | 0 | 234
  Week 4 of of cycle 3 - Urea nitrogen (mmol/L) |  |  | 0.01 (1.272)
  Week 4 of of cycle 4 - Cholesterol (mmol/L): number analyzed (Participants) | 0 | 0 | 127
  Week 4 of of cycle 4 - Cholesterol (mmol/L) |  |  | 0.040 (0.6614)
  Week 4 of of cycle 4 - Glucose (mmol/L): number analyzed (Participants) | 0 | 0 | 127
  Week 4 of of cycle 4 - Glucose (mmol/L) |  |  | -0.098 (1.9131)
  Week 4 of of cycle 4 - Potassium (mmol/L): number analyzed (Participants) | 0 | 0 | 127
  Week 4 of of cycle 4 - Potassium (mmol/L) |  |  | 0.08 (0.039)
  Week 4 of of cycle 4 - Sodium (mmol/L): number analyzed (Participants) | 0 | 0 | 127
  Week 4 of of cycle 4 - Sodium (mmol/L) |  |  | 0.2 (1.87)
  Week 4 of of cycle 4 - Urea nitrogen (mmol/L): number analyzed (Participants) | 0 | 0 | 127
  Week 4 of of cycle 4 - Urea nitrogen (mmol/L) |  |  | 0.06 (1.398)

20. Secondary Outcome: Change From to Baseline of Bilirubin, Creatinin
Description: Safety assessments by evaluating change from baseline of Bilirubin, Creatinin as per the study schedule
Time Frame: as for outcome 10
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: μmol/L
Arm/Group | Botulinum Toxin A | Placebo | Botulinum Toxin A Open Label Extension Arm
Number analyzed (Participants) | 259 | 84 | 301
μmol/L
  Week 4 of cycle 1 - Bilirubin (μmol/L): number analyzed (Participants) | 254 | 82 | 0
  Week 4 of cycle 1 - Bilirubin (μmol/L) | 0.05 (3.555) | -0.14 (3.597) |
  Week 4 of cycle 1 - Creatinine (μmol/L): number analyzed (Participants) | 259 | 84 | 0
  Week 4 of cycle 1 - Creatinine (μmol/L) | 0.52 (8.404) | -0.30 (6.556) |
  Week 4 of cycle 2 - Bilirubin (μmol/L): number analyzed (Participants) | 0 | 0 | 300
  Week 4 of cycle 2 - Bilirubin (μmol/L) |  |  | -0.12 (3.329)
  Week 4 of cycle 2 - Creatinine (μmol/L): number analyzed (Participants) | 0 | 0 | 301
  Week 4 of cycle 2 - Creatinine (μmol/L) |  |  | -0.49 (8.550)
  Week 4 of cycle 3 - Bilirubin (μmol/L): number analyzed (Participants) | 0 | 0 | 233
  Week 4 of cycle 3 - Bilirubin (μmol/L) |  |  | -0.14 (3.283)
  Week 4 of cycle 3 - Creatinine (μmol/L): number analyzed (Participants) | 0 | 0 | 234
  Week 4 of cycle 3 - Creatinine (μmol/L) |  |  | 0.06 (9.553)
  Week 4 of cycle 4 - Bilirubin (μmol/L): number analyzed (Participants) | 0 | 0 | 127
  Week 4 of cycle 4 - Bilirubin (μmol/L) |  |  | 0.52 (3.203)
  Week 4 of cycle 4 - Creatinine (μmol/L): number analyzed (Participants) | 0 | 0 | 127
  Week 4 of cycle 4 - Creatinine (μmol/L) |  |  | -0.66 (9.536)

21. Secondary Outcome: Change From Baseline of Erythrocytes
Description: Safety assessments by evaluating change from baseline of Erythrocytes as per the study schedule
Time Frame: as for outcome 10
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: x10^12 cells/L
Arm/Group | Botulinum Toxin A | Placebo | Botulinum Toxin A Open Label Extension Arm
Number analyzed (Participants) | 250 | 82 | 299
x10^12 cells/L
  Cycle 1: number analyzed (Participants) | 250 | 82 | 0
  Cycle 1 | -0.002 (0.2425) | -0.038 (0.2194) |
  Cycle 2: number analyzed (Participants) | 0 | 0 | 299
  Cycle 2 |  |  | 0.032 (0.2091)
  Cycle 3: number analyzed (Participants) | 0 | 0 | 234
  Cycle 3 |  |  | 0.063 (0.2619)
  Cycle 4: number analyzed (Participants) | 0 | 0 | 126
  Cycle 4 |  |  | 0.041 (0.2716)

22. Secondary Outcome: Change From Baseline of Erythrocytes MCV
Description: Safety assessments by evaluating change from baseline of Erythrocytes MCV as per the study schedule
Time Frame: as for outcome 10
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: fL
Arm/Group | Botulinum Toxin A | Placebo | Botulinum Toxin A Open Label Extension Arm
Number analyzed (Participants) | 250 | 82 | 299
fL
  Cycle 1: number analyzed (Participants) | 250 | 82 | 0
  Cycle 1 | -0.78 (2.615) | -0.79 (2.860) |
  Cycle 2: number analyzed (Participants) | 0 | 0 | 299
  Cycle 2 |  |  | -0.38 (3.070)
  Cycle 3: number analyzed (Participants) | 0 | 0 | 234
  Cycle 3 |  |  | 0.53 (4.209)
  Cycle 4: number analyzed (Participants) | 0 | 0 | 126
  Cycle 4 |  |  | 2.18 (3.875)

23. Secondary Outcome: Change From Baseline of Erythrocyte MCHC, Hemoglobin
Description: Safety assessments by evaluating change from baseline of Erythrocyte MCHC, Hemoglobin as per the study schedule
Time Frame: as for outcome 10
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | Botulinum Toxin A | Placebo | Botulinum Toxin A Open Label Extension Arm
Number analyzed (Participants) | 250 | 82 | 299
g/dL
  Week 4 of cycle 1 - Erythrocyte MCHC (g/dL): number analyzed (Participants) | 250 | 82 | 0
  Week 4 of cycle 1 - Erythrocyte MCHC (g/dL) | 0.32 (0.954) | 0.33 (1.041) |
  Week 4 of cycle 1 - Hemoglobin (g/dL): number analyzed (Participants) | 250 | 82 | 0
  Week 4 of cycle 1 - Hemoglobin (g/dL) | 0.02 (0.732) | -0.09 (0.740) |
  Week 4 of cycle 2 - Erythrocyte MCHC (g/dL): number analyzed (Participants) | 0 | 0 | 299
  Week 4 of cycle 2 - Erythrocyte MCHC (g/dL) |  |  | 0.16 (1.070)
  Week 4 of cycle 2 - Hemoglobin (g/dL): number analyzed (Participants) | 0 | 0 | 299
  Week 4 of cycle 2 - Hemoglobin (g/dL) |  |  | 0.12 (0.638)
  Week 4 of cycle 3 - Erythrocyte MCHC (g/dL): number analyzed (Participants) | 0 | 0 | 234
  Week 4 of cycle 3 - Erythrocyte MCHC (g/dL) |  |  | -0.12 (1.366)
  Week 4 of cycle 3 - Hemoglobin (g/dL): number analyzed (Participants) | 0 | 0 | 234
  Week 4 of cycle 3 - Hemoglobin (g/dL) |  |  | -0.21 (0.821)
  Week 4 of cycle 4 - Erythrocyte MCHC (g/dL): number analyzed (Participants) | 0 | 0 | 126
  Week 4 of cycle 4 - Erythrocyte MCHC (g/dL) |  |  | -0.65 (1.306)
  Week 4 of cycle 4 - Hemoglobin (g/dL): number analyzed (Participants) | 0 | 0 | 126
  Week 4 of cycle 4 - Hemoglobin (g/dL) |  |  | -0.15 (0.921)

24. Secondary Outcome: Change From Baseline of Lymphocytes/Leukocytes, Monocytes/Leukocytes, Neutrophils/Leukocytes, Basophiles/Leukocytes, Eosinophils/Leukocytes
Description: Safety assessments by evaluating change from baseline of Lymphocytes/leukocytes, Monocytes/leukocytes, Neutrophils/leukocytes, Basophiles/leukocytes, Eosinophils/leukocytes as per the study schedule
Time Frame: as for outcome 10
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: % of leukocytes
Arm/Group | Botulinum Toxin A | Placebo | Botulinum Toxin A Open Label Extension Arm
Number analyzed (Participants) | 250 | 82 | 299
% of leukocytes
  Week 4 of cycle 1 - Basophiles/leukocytes (%): number analyzed (Participants) | 250 | 82 | 0
  Week 4 of cycle 1 - Basophiles/leukocytes (%) | 0.05 (0.669) | 0.14 (0.890) |
  Week 4 of cycle 1 - Eosinophils/leukocytes (%): number analyzed (Participants) | 250 | 82 | 0
  Week 4 of cycle 1 - Eosinophils/leukocytes (%) | 0.14 (1.090) | 0.05 (1.292) |
  Week 4 of cycle 1 - Lymphocytes/leukocytes (%): number analyzed (Participants) | 250 | 82 | 0
  Week 4 of cycle 1 - Lymphocytes/leukocytes (%) | -0.26 (6.724) | -1.13 (5.468) |
  Week 4 of cycle 1 - Monocytes/leukocytes (%): number analyzed (Participants) | 250 | 82 | 0
  Week 4 of cycle 1 - Monocytes/leukocytes (%) | -0.40 (2.337) | -0.48 (2.350) |
  Week 4 of cycle 1 - Neutrophils/leukocytes (%): number analyzed (Participants) | 250 | 82 | 0
  Week 4 of cycle 1 - Neutrophils/leukocytes (%) | 0.47 (7.610) | 1.41 (6.219) |
  Week 4 of cycle 2 - Basophiles/leukocytes (%): number analyzed (Participants) | 0 | 0 | 299
  Week 4 of cycle 2 - Basophiles/leukocytes (%) |  |  | -0.04 (0.837)
  Week 4 of cycle 2 - Eosinophils/leukocytes (%): number analyzed (Participants) | 0 | 0 | 299
  Week 4 of cycle 2 - Eosinophils/leukocytes (%) |  |  | 0.13 (1.554)
  Week 4 of cycle 2 - Lymphocytes/leukocytes (%): number analyzed (Participants) | 0 | 0 | 299
  Week 4 of cycle 2 - Lymphocytes/leukocytes (%) |  |  | 0.80 (6.802)
  Week 4 of cycle 2 - Monocytes/leukocytes (%): number analyzed (Participants) | 0 | 0 | 299
  Week 4 of cycle 2 - Monocytes/leukocytes (%) |  |  | -0.04 (1.559)
  Week 4 of cycle 2 - Neutrophils/leukocytes (%): number analyzed (Participants) | 0 | 0 | 299
  Week 4 of cycle 2 - Neutrophils/leukocytes (%) |  |  | -0.84 (7.660)
  Week 4 of cycle 3 - Basophiles/leukocytes (%): number analyzed (Participants) | 0 | 0 | 234
  Week 4 of cycle 3 - Basophiles/leukocytes (%) |  |  | -0.25 (0.764)
  Week 4 of cycle 3 - Eosinophils/leukocytes (%): number analyzed (Participants) | 0 | 0 | 234
  Week 4 of cycle 3 - Eosinophils/leukocytes (%) |  |  | 0.06 (1.788)
  Week 4 of cycle 3 - Lymphocytes/leukocytes (%): number analyzed (Participants) | 0 | 0 | 234
  Week 4 of cycle 3 - Lymphocytes/leukocytes (%) |  |  | 0.82 (7.814)
  Week 4 of cycle 3 - Monocytes/leukocytes (%): number analyzed (Participants) | 0 | 0 | 234
  Week 4 of cycle 3 - Monocytes/leukocytes (%) |  |  | -0.16 (1.790)
  Week 4 of cycle 3 - Neutrophils/leukocytes (%): number analyzed (Participants) | 0 | 0 | 234
  Week 4 of cycle 3 - Neutrophils/leukocytes (%) |  |  | -0.47 (9.240)
  Week 4 of cycle 4 - Basophiles/leukocytes (%): number analyzed (Participants) | 0 | 0 | 126
  Week 4 of cycle 4 - Basophiles/leukocytes (%) |  |  | -0.23 (0.663)
  Week 4 of cycle 4 - Eosinophils/leukocytes (%): number analyzed (Participants) | 0 | 0 | 126
  Week 4 of cycle 4 - Eosinophils/leukocytes (%) |  |  | -0.26 (1.191)
  Week 4 of cycle 4 - Lymphocytes/leukocytes (%): number analyzed (Participants) | 0 | 0 | 126
  Week 4 of cycle 4 - Lymphocytes/leukocytes (%) |  |  | 1.68 (6.869)
  Week 4 of cycle 4 - Monocytes/leukocytes (%): number analyzed (Participants) | 0 | 0 | 126
  Week 4 of cycle 4 - Monocytes/leukocytes (%) |  |  | 0.06 (2.434)
  Week 4 of cycle 4 - Neutrophils/leukocytes (%): number analyzed (Participants) | 0 | 0 | 126
  Week 4 of cycle 4 - Neutrophils/leukocytes (%) |  |  | -1.34 (7.460)

25. Secondary Outcome: Change From Baseline of Systolic and Diastolic Blood Pressure
Description: Safety assessments by evaluating change from baseline of Systolic and Diastolic Blood Pressure as per the study schedule
Time Frame: as for outcome 10
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Botulinum Toxin A | Placebo | Botulinum Toxin A Open Label Extension Arm
Number analyzed (Participants) | 263 | 85 | 305
mmHg
  Week 4 of cycle 1 - Systolic Blood Pressure (mmHg): number analyzed (Participants) | 263 | 85 | 0
  Week 4 of cycle 1 - Systolic Blood Pressure (mmHg) | -0.7 (11.13) | -0.2 (10.50) |
  Week 4 of cycle 1 - Diastolic Blood Pressure (mmHg): number analyzed (Participants) | 263 | 85 | 0
  Week 4 of cycle 1 - Diastolic Blood Pressure (mmHg) | -1.0 (7.54) | 1.3 (8.16) |
  Week 4 of cycle 2 - Systolic Blood Pressure (mmHg): number analyzed (Participants) | 0 | 0 | 305
  Week 4 of cycle 2 - Systolic Blood Pressure (mmHg) |  |  | -0.9 (11.66)
  Week 4 of cycle 2 - Diastolic Blood Pressure (mmHg): number analyzed (Participants) | 0 | 0 | 305
  Week 4 of cycle 2 - Diastolic Blood Pressure (mmHg) |  |  | 0.0 (7.79)
  Week 4 of cycle 3 - Systolic Blood Pressure (mmHg): number analyzed (Participants) | 0 | 0 | 235
  Week 4 of cycle 3 - Systolic Blood Pressure (mmHg) |  |  | -1.7 (12.06)
  Week 4 of cycle 3 - Diastolic Blood Pressure (mmHg): number analyzed (Participants) | 0 | 0 | 235
  Week 4 of cycle 3 - Diastolic Blood Pressure (mmHg) |  |  | -0.4 (8.02)
  Week 4 of cycle 4 - Systolic Blood Pressure (mmHg): number analyzed (Participants) | 0 | 0 | 128
  Week 4 of cycle 4 - Systolic Blood Pressure (mmHg) |  |  | -1.8 (13.40)
  Week 4 of cycle 4 - Diastolic Blood Pressure (mmHg): number analyzed (Participants) | 0 | 0 | 128
  Week 4 of cycle 4 - Diastolic Blood Pressure (mmHg) |  |  | -0.2 (7.38)

26. Secondary Outcome: Change From Baseline of Pulse Rate
Description: Safety assessments by evaluating change from baseline of Pulse rate as per the study schedule
Time Frame: as for outcome 10
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: bpm
Arm/Group | Botulinum Toxin A | Placebo | Botulinum Toxin A Open Label Extension Arm
Number analyzed (Participants) | 263 | 85 | 305
bpm
  Cycle 1: number analyzed (Participants) | 263 | 85 | 0
  Cycle 1 | -1.7 (10.83) | 0.1 (10.24) |
  Cycle 2: number analyzed (Participants) | 0 | 0 | 305
  Cycle 2 |  |  | 1.2 (9.11)
  Cycle 3: number analyzed (Participants) | 0 | 0 | 235
  Cycle 3 |  |  | 2.2 (10.73)
  Cycle 4: number analyzed (Participants) | 0 | 0 | 128
  Cycle 4 |  |  | 0.7 (10.73)

27. Secondary Outcome: Number of Participants With Normal and Abnormal Electrocardiogram
Description: Safety assessments by evaluating Electrocardiogram as per the study schedule
Time Frame: Week 4 and last visit of Treatment Cycle 1 (End of Cycle procedures), conducted upon confirmation of eligibility for retreatment, assessed starting 12 weeks post-treatment with 4-weekly evaluations up to a max. of 48 weeks post treatment.
Population: The population used consists of all subjects who received at least one injection with study medication and who have data available for the respective visit and category of baseline electrocardiogram interpretation. Participants were analyzed as treated.
Measure: Count of Participants; unit: Participants
Groups:
- Botulinum Toxin A - Normal Baseline Electrocardiogram Interpretation: Botulinum Toxin A will be administered in double blind fashion in Treatment Cycle 1. 20 Units will be administered (divided in five 0.1 mL i.m injections) into glabellar area.
  Botulinum Toxin A: Injection, 20 Units divided in five 0.1 mL i.m injections into the glabellar area
  Subjects had an electrocardiogram interpretation of normal at baseline.
- Botulinum Toxin A - Abnormal Baseline Electrocardiogram Interpretation: Botulinum Toxin A will be administered in double blind fashion in Treatment Cycle 1. 20 Units will be administered (divided in five 0.1 mL i.m injections) into glabellar area.
  Botulinum Toxin A: Injection, 20 Units divided in five 0.1 mL i.m injections into the glabellar area
  Subjects had an electrocardiogram interpretation of abnormal at baseline.
- Placebo - Normal Baseline Electrocardiogram Interpretation: Placebo will be administered in double blind fashion in Treatment Cycle 1 divided in five 0.1 mL injections into the glabellar area.
  Placebo: injection, sodium chloride 0.9 % divided in five 0.1 mL i.m injections into the glabellar area
  Subjects had an electrocardiogram interpretation of normal at baseline.
- Placebo - Abnormal Baseline Electrocardiogram Interpretation: Placebo will be administered in double blind fashion in Treatment Cycle 1 divided in five 0.1 mL injections into the glabellar area.
  Placebo: injection, sodium chloride 0.9 % divided in five 0.1 mL i.m injections into the glabellar area
  Subjects had an electrocardiogram interpretation of abnormal at baseline.
Arm/Group | Botulinum Toxin A - Normal Baseline Electrocardiogram Interpretation | Botulinum Toxin A - Abnormal Baseline Electrocardiogram Interpretation | Placebo - Normal Baseline Electrocardiogram Interpretation | Placebo - Abnormal Baseline Electrocardiogram Interpretation
Number analyzed (Participants) | 238 | 28 | 77 | 12
Participants
  Cycle 1 Week 4 - Electrocardiogram Interpretation: number analyzed (Participants) | 236 | 27 | 74 | 11
  Cycle 1 Week 4 - Electrocardiogram Interpretation: Normal | 223 | 5 | 71 | 3
  Cycle 1 Week 4 - Electrocardiogram Interpretation: Abnormal | 13 | 22 | 3 | 8
  Cycle 1 End of Cycle Visit - Electrocardiogram Interpretation: number analyzed (Participants) | 208 | 25 | 73 | 11
  Cycle 1 End of Cycle Visit - Electrocardiogram Interpretation: Normal | 198 | 6 | 69 | 3
  Cycle 1 End of Cycle Visit - Electrocardiogram Interpretation: Abnormal | 10 | 19 | 4 | 8

ADVERSE EVENTS:
Time Frame: Up to 60 weeks post first treatment
Arm/Group | Botulinum Toxin A | Placebo | Botulinum Toxin A Open Label Extension Arm
All-Cause Mortality (participants affected / at risk) | 0/266 | 0/89 | 0/323
Serious Adverse Events (participants affected / at risk) | 1/266 | 1/89 | 4/323
Other Adverse Events (participants affected / at risk) | 12/266 | 6/89 | 14/323
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Botulinum Toxin A (N=266) | Placebo (N=89) | Botulinum Toxin A Open Label Extension Arm (N=323)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Goitre (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
Foot deformity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Botulinum Toxin A (N=266) | Placebo (N=89) | Botulinum Toxin A Open Label Extension Arm (N=323)
Nasopharyngitis (Infections and infestations) | 2 (2) | 3 (3) | 9 (9)
Tooth fracture (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 1 (1)
Headache (Nervous system disorders) | 10 (10) | 2 (2) | 5 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2019-07-15): https://cdn.clinicaltrials.gov/large-docs/82/NCT03985982/Prot_000.pdf
  • Statistical Analysis Plan (2020-11-04): https://cdn.clinicaltrials.gov/large-docs/82/NCT03985982/SAP_001.pdf